CLINICAL TRIAL: NCT00145080
Title: Evaluation of Strategies for Increasing Osteoporosis Screening and Treatment in a Managed Care Organization
Brief Title: Comparison of Osteoporosis Disease Management Strategies (0000-039)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0000-039; 039; 2005_050
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Behavioral: Disease Management Assessment

SUMMARY:
The purpose of this study is to assess the impact of disease management interventions on bone mineral density screening rates and osteoporosis treatment rates in women age 50-64 years at high risk for osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Members of the Harvard Pilgrim Health Plan

Exclusion Criteria:

* Individuals who are not members of the Harvard Pilgrim Health Plan

Ages: 50 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4685 (Actual)
Dates: Start 2004-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density screening rates

SECONDARY OUTCOMES:
Medications adoptions; Medications adherence

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Heyworth L, Kleinman K, Oddleifson S, Bernstein L, Frampton J, Lehrer M, Salvato K, Weiss TW, Simon SR, Connelly M. Comparison of interactive voice response, patient mailing, and mailed registry to encourage screening for osteoporosis: a randomized controlled trial. Osteoporos Int. 2014 May;25(5):1519-26. doi: 10.1007/s00198-014-2629-1. Epub 2014 Feb 25. PMID 24566584